CLINICAL TRIAL: NCT02292550
Title: A Phase Ib/II Study of the ALK Inhibitor Ceritinib in Combination With the CDK4/6 Inhibitor LEE011 in Patients With ALK-positive Non-Small Cell Lung Cancer
Brief Title: Study of Safety and Efficacy of LEE011 and Ceritinib in Patients With ALK-positive Non-small Cell Lung Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011X2110C
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2019-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; ALK translocation; ALK-positive; NSCLC; LEE011; CDK4/6 inhibitor; EML4-ALK; cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — ribociclib; ceritinib

STUDY DESIGN:
Intervention Model Description: This was a multi-center, open-label, dose finding, Phase Ib dose escalation study to estimate the maximum tolerated doses (MTD(s))
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Ribociclib 100 mg + Ceritinib 300 mg (Experimental): LEE011 capsule for oral use (ribociclib) and Ceritinib for oral use
  Interventions: Drug: Ribociclib; Drug: Ceritinib
- Ribociclib 100 mg + Ceritinib 450 mg (Experimental): LEE011 capsule for oral use (ribociclib) and Ceritinib for oral use
  Interventions: Drug: Ribociclib; Drug: Ceritinib
- Ribociclib 200 mg + Ceritinib 300 mg (Experimental): LEE011 capsule for oral use (ribociclib) and Ceritinib for oral use
  Interventions: Drug: Ribociclib; Drug: Ceritinib
- Ribociclib 200 mg + Ceritinib 450 mg (Experimental): LEE011 capsule for oral use (ribociclib) and Ceritinib for oral use
  Interventions: Drug: Ribociclib; Drug: Ceritinib
- Ribociclib 300 mg + Ceritinib 450 mg (Experimental): LEE011 capsule for oral use (ribociclib) and Ceritinib for oral use
  Interventions: Drug: Ribociclib; Drug: Ceritinib

INTERVENTIONS:
Drug: Ribociclib — CDK 4/6 inhibitor
  Other Names: LEE011
Drug: Ceritinib — ALK inhibitor
  Other Names: LDK378, Zykadia

SUMMARY:
This was a Phase Ib/II study of the ALK inhibitor ceritinib in combination with the CDK4/6 inhibitor LEE011 in patients with ALK-positive non-small cell lung cancer.

The purpose of the study was to determine the MTD/RP2D of the LEE011 and ceritinib combination and evaluate whether the combination was safe and had beneficial effects in ALK-positive advanced non-small cell lung cancer patients.

This trial did not progress to Phase II. Trial population terminated before reaching Phase II

DETAILED DESCRIPTION:
In Sep-2016, Novartis made a decision not to move into phase ll after the primary objective for this study was met. Because the study never made it to phase ll, the study phase has been changed from a phase l/ll to a phase l.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with ALK-positive advanced NSCLC. The tumor must be ALK-positive as determined by ALK rearrangement in ≥15% of cells (as measured by FISH using the Vysis break-apart ALK probe) or by using the Ventana ALK IHC test. The analysis may be performed locally.
* Eastern cooperative oncology group (ECOG) performance status ≤ 2.
* Measurable disease as per RECIST v1.1
* Availability of tumor sample:

For ALK inhibitor naïve patients:

o A representative tumor sample must be submitted. An archival tumor specimen is acceptable

For patients after progression on an ALK inhibitor:

o A new tumor biopsy is required unless a biopsy performed after progression on the patient's most recent ALK inhibitor is available for submission For all patients a newly obtained tumor specimen must be submitted if no appropriate archival sample is available. In the event that no sample is available and a new biopsy cannot be obtained, enrollment may be considered after discussion with the sponsor.

Exclusion Criteria:

* For Phase I part:

  o Patients who have not previously received at least one line of therapy for ALK-positive NSCLC
* For Phase II part:

  * Group A: prior therapy with any ALK inhibitor is not permitted.
  * Group B: progression following any ALK inhibitor(s) other than ceritinib is required and the last dose of the ALK inhibitor must be no more than 60 days prior to the first dose of study drug. Prior ceritinib is not permitted.
  * Group C: progression following ceritinib is required and the last dose of ceritinib must be no more than 60 days prior to the first dose of study drug.
* Patients who have previously been unable to tolerate ceritinib, in the opinion of the investigator. Exceptions to this exclusion include nausea, vomiting and diarrhea in patients taking ceritinib under fasted conditions.
* Patients with symptomatic central nervous system (CNS) metastases who are neurologically unstable or require increasing doses of steroids or local CNS-directed therapy to control their CNS disease
* Patients with abnormal laboratory values during screening and on day 1 of pre-dose
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of ceritinib or LEE011
* Patients who are currently receiving treatment (that cannot be discontinued at least 1 week prior to the initiation of the study) with agents that are known to be any of the following: strong inducers or inhibitors of CYP3A4/5; sensitive substrates of CYP3A; substrates of CYP3A4/5 or CYP2C9 with a narrow therapeutic index.
* Patient has a history of pancreatitis or history of increased amylase or lipase that was due to pancreatic disease.
* Patient with impaired cardiac function or any clinically significant uncontrolled cardiac disease, and/or, cardiac repolarization abnormality, including any of the following:

Clinically significant heart disease such as CHF requiring treatment (NYH grade ≥ 2), history of angina pectoris, myocardial infarction, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to study entry, documented cardiomyopathy, or left ventricular ejection fraction (LVEF) < 50% as determined by multiple gated acquisition scan (MUGA) or echocardiogram (ECHO).

Uncontrolled systolic blood pressure (SBP) ≥160 mmHg and/or diastolic blood pressure (DBP) ≥100 mmHg, with or without anti-hypertensive medication. Initiation or adjustment of antihypertensive medication (s) is allowed prior to screening, Systolic blood pressure (SBP) <90 mmHg Standard 12-lead ECG values defined as the mean of the triplicate ECGs and assessed by central laboratory

* QTcF interval at screening >450 msec (using Fridericia's correction)
* Resting heart rate <50 bpm or > 90 bpm

Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

* Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia
* Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued or replaced by safe alternative medication (e.g. within 5 half-lives or 7 days prior to starting study drug)
* Inability to determine the QTcF interval Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third degree AV block).

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Incidence rate of dose limiting toxicities (DLTs) during the first cycle of treatment (Phase Ib ) | 1 month
  Maximum Tolerated Dose(s) (MTD(s)) and/or recommended phase 2 dose (RP2D(s)) and schedule of LEE011 in combination with ceritinib in ALK-positive non-small cell lung cancer (NSCLC) patients.
  Cycle = 28 days
Overall Response Rate (ORR) as per RECIST v1.1 | Up to 24 months
  Preliminary anti-tumor activity of the LEE011 and ceritinib combination
Exposure to LEE011 and ceritinib (Phase Ib ) | Up to 6 months
  Measurement of pharmacokinetics (PK) parameters (AUC0-24h at C1D15)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) - Phase Ib & II | Up to 24 months
  Preliminary measure of anti-tumor activity of LEE011 and ceritinib combination
Frequency of adverse events/serious adverse events | Up to 24 months
  Characterization of the safety and tolerability of the LEE011 and ceritinib combination as determined by changes in laboratory values and electrocardiograms
PK parameters of LEE011 and ceritinib | Up to 6 months
  Characterization of the PK of LEE011 and ceritinib
Frequency of dose interruptions and dose reductions (phase lb & ll) | Up to 24 months
  Characterization of tolerability
Progression free survival (PFS) per RECIST v1.1 - Phase Ib & II | Up to 24 months
  Preliminary measures of anti-tumor activity of LEE011 and ceritinib combination
Duration of response (DOR) | Up to 24 months
  Preliminary measure of anti-tumor activity of LEE011 and ceritinib combination
Time to response (TTR) - Phase Ib & II | Up to 24 months
  Preliminary measures of anti-tumor activity of LEE011 and ceritinib combination
Disease Control Rate (DCR) - Phase Ib & II | Up to 24 months
  Preliminary measures of anti-tumor activity of LEE011 and ceritinib combination
Overall survival (OS) - Phase Ib & II | Up to 24 months
  Preliminary measures of anti-tumor activity of LEE011 and ceritinib combination
Severity of adverse events/serious adverse events | Up to 24 months
  Characterization of the safety and tolerability of the LEE011 and ceritinib combination as determined by changes in laboratory values and electrocardiograms.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Novartis Investigative Site, Boston, Massachusetts, United States
- Novartis Investigative Site, Marseille, France
- Italy (2):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Rozzano, MI
- Novartis Investigative Site, Seoul, Seocho Gu, South Korea
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Taiwan (2):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Taipei

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Results for CLEE011X2110C can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17544